CLINICAL TRIAL: NCT03983993
Title: A Phase II Study of Niraparib in Combination With EGFR Inhibitor Panitumumab in Patients With Advanced Colorectal Cancer
Brief Title: Niraparib and Panitumumab in Patients With Advanced or Metastatic Colorectal Cancer
Acronym: NIPAVect
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: GlaxoSmithKline (Industry); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Olatunji Alese, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00107377; NCI-2018-02757 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4517-18 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Advanced Microsatellite Stable Colorectal Carcinoma; Metastatic Microsatellite Stable Colorectal Carcinoma; Microsatellite Stable; RAS Wild Type; Stage IV Colorectal Cancer AJCC v8; MSI-H Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — niraparib; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (niraparib, panitumumab) (Experimental): Patients receive 200 or 300 mg niraparib orally once daily on days 1-28 and 6 mg/kg panitumumab intravenously over 60-90 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Niraparib; Biological: Panitumumab

INTERVENTIONS:
Drug: Niraparib — Given PO
  Other Names: MK-4827; Zejula
Biological: Panitumumab — Given IV
  Other Names: ABX-EGF; Vectibix

SUMMARY:
This phase II trial studies the side effects and how well niraparib and panitumumab work in treating patients with colorectal cancer that has spread to other places in the body. Niraparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as panitumumab, may help the body's immune system attack the cancer and may interfere with the ability of tumor cells to grow and spread. Giving niraparib and panitumumab may work better in treating patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the activity of the combination of niraparib with epidermal growth factor receptor (EGFR) inhibitor panitumumab in previously treated patients with rat sarcoma gene (RAS) wild type (WT) metastatic colorectal cancer.

SECONDARY OBJECTIVES:

I. Define the toxicity profile of the combination of niraparib and panitumumab.

II. Evaluate the activity of the combination of niraparib and panitumumab in previously treated patients with metastatic colorectal cancer.

OUTLINE:

Patients receive niraparib orally (PO) once daily (QD) on days 1-28 and panitumumab intravenously (IV) over 60-90 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 6 months for 2 years, and then annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have advanced, metastatic RAS wildtype colorectal cancer and must have received at least one line of systemic therapy. Both microsatellite (MSI) high and stable (MSS) patients are eligible
* Participants may have been intolerant of, progressed on, or failed at least one line of systemic chemotherapy. Patients who are currently on first line Oxaliplatin-containing chemotherapy regimen are allowed on the trial if they have remained stable or better ([partial response]PR or [complete response]CR) for at least 4 months on that line of treatment and are being considered for maintenance therapy as standard of care
* Histologic or cytologic diagnosis of colorectal cancer
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
* Absolute neutrophil count ≥ 1,500/µL
* Platelets ≥ 100,000/µL
* Hemoglobin ≥ 9 g/dL
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault equation
* Total bilirubin ≤ 1.5 x ULN (≤ 2.0 in patients with known Gilberts syndrome) OR direct bilirubin ≤ 1 x ULN
* Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
* Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment
* Female participant has a negative urine or serum pregnancy test within 7 days prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 180 days after the last dose of study
* Male participant agrees to use an adequate method of contraception starting with the first dose of study treatment through 180 days after the last dose of study treatment
* Participant must be able to provide written informed consent

Exclusion Criteria:

* Participant must not be simultaneously enrolled in any interventional clinical trial
* Prior therapy with poly ADP (adenosine diphosphate) ribose polymerase (PARP) inhibitors or with EGFR inhibitors approved for the treatment of colorectal cancer (cetuximab or panitumumab)
* Patients with a history of interstitial pneumonitis or pulmonary fibrosis, or evidence of interstitial pneumonitis or pulmonary fibrosis during screening
* Inability to take oral medications
* Participant has had radiation therapy encompassing > 20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to day 1 of protocol therapy
* Participant must not have a known hypersensitivity to components or excipients of niraparib or panitumumab
* Participant must not have a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Participant must not have had diagnosis, detection, or treatment of another type of cancer ≤ 2 years prior to initiating protocol therapy (except basal or squamous cell carcinoma of the skin and cervical cancer that has been definitively treated)
* Participant must not have known active, symptomatic brain or leptomeningeal metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2026-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Olatunji Alese, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Niraparib, Panitumumab)
Started | 25
Completed | 24
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Niraparib, Panitumumab)
Number analyzed (Participants) | 25
Age, Continuous [Median (Standard Deviation); unit: years] | 58.5 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR)
Description: The efficacy, as measured by clinical benefit rate (CBR), will be assessed for the total number of patients enrolled. CBR = (Complete Response + Partial Response + Stable Disease [CR +PR + SD] rate. Response will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 criteria using an independent review.
Time Frame: 3 years and 7 months post treatment
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Niraparib, Panitumumab)
Number analyzed (Participants) | 24
percentage of participants | 83.3

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) is defined as the percentage of patients with complete response (CR) or partial response (PR), as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 criteria using an independent review.
Time Frame: Up to 5 years post treatment
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Niraparib, Panitumumab)
Number analyzed (Participants) | 24
percentage of participants | 25

3. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) is defined as the time from the initial response (complete response [CR] or partial response [PR]) until the time of first documentation of disease progression, as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 criteria using an independent review.
Time Frame: Up to 5 years post treatment
Reporting Status: Not Posted

4. Secondary Outcome: Progression Free Survival (PFS)
Description: For progression free survival (PFS), progression or death from any cause will be defined as the event. Progression will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 criteria using an independent review. Patients will be censored at time of last follow-up.
Time Frame: Up to 5 years post treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Niraparib, Panitumumab)
Number analyzed (Participants) | 24
months | 5.6 [3.7 to 6.9]

5. Secondary Outcome: Overall Survival (OS)
Description: For overall survival (OS), death from any cause will be defined as the event. Patients will be censored at time of last follow-up.
Time Frame: Up to 5 years post treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Niraparib, Panitumumab)
Number analyzed (Participants) | 24
months | 20.9 [9.2 to NA] — Median Overall Survival- 20.9 months (95% CI: 9.2, NR). The NA means the upper bound of 95%CI of median OS is not estimatable by Kaplan-Meier method due to not having a sufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: 5 years after study enrollment
Arm/Group | Treatment (Niraparib, Panitumumab)
All-Cause Mortality (participants affected / at risk) | 10/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 17/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Niraparib, Panitumumab) (N=24)
Rash (Skin and subcutaneous tissue disorders) | 17
Anemia (Blood and lymphatic system disorders) | 8
Fatigue (General disorders) | 8
Constipation (Gastrointestinal disorders) | 7
Aspartate aminotransferase increased (Investigations) | 5
Hypokalemia (Investigations) | 5
Oral mucositis (Gastrointestinal disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Alkaline Phosphatase increased (Investigations) | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 3
Hyponatremia (Investigations) | 3
Nail changes (Skin and subcutaneous tissue disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 2
Elevated bilirubin (Hepatobiliary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dizziness (Nervous system disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Fever (Infections and infestations) | 2
Purpura (Skin and subcutaneous tissue disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Weight loss (Gastrointestinal disorders) | 2
Sore throat (Gastrointestinal disorders) | 2
Gastroesophageal reflux (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/93/NCT03983993/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/93/NCT03983993/ICF_000.pdf